CLINICAL TRIAL: NCT02745964
Title: A Comparison of LMA-Supreme and I-gel for the Incidence of Postoperative Sore Throat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was closed earlier than planned because of lack of research staff.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2016-0144
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA supreme (Experimental): Anesthesia is maintained using LMA supreme during surgery.
  Interventions: Device: LMA supreme
- I-gel (Active Comparator): Anesthesia is maintained using I-gel during surgery.
  Interventions: Device: I-gel

INTERVENTIONS:
Device: LMA supreme — Anesthesia is maintained using LMA supreme in LMA supreme group or using I-gel in I-gel group according to the randomly allocated groups.
  Arms: LMA supreme
Device: I-gel — Anesthesia is maintained using LMA supreme in LMA supreme group or using I-gel in I-gel group according to the randomly allocated groups.
  Arms: I-gel

SUMMARY:
The purpose of this study is to investigate and compare the incidence of the postoperative sore throat between LMA supreme and I-gel.

ELIGIBILITY:
Inclusion Criteria:

- adult patients aged over 19 years who are scheduled for elective surgery under general anesthesia using the laryngeal mask airway

Exclusion Criteria:

* Anticipated difficult airway
* Expected duration of surgery more than 4 hours
* body mass index more than 35 kg/m2
* pregnancy
* Upper gastrointestinal surgery or open abdominal surgery.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2016-06-11 (Actual); Study Completion 2016-06-11 (Actual)

PRIMARY OUTCOMES:
Postoperative sore throat | within 24 hours after the end of surgery.
  The postoperative sore throat will be evaluated after the end of surgery by the investigator who are blinded to the group assignments. The investigator will ask the participant about his/her sore throat status.

SECONDARY OUTCOMES:
Postoperative dysphagia | within 24 hours after the end of surgery
  The postoperative dysphagia will be evaluated after the end of surgery by the investigator who are blinded to the group assignments. The investigator will ask the participant about his/her status.
Postoperative dysphonia | within 24 hours after the end of surgery
  The postoperative dysphonia will be evaluated after the end of surgery by the investigator who are blinded to the group assignments. The investigator will ask the participant about his/her status.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain MedicineSeverance Hospital, Yonsei University Health System, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data